CLINICAL TRIAL: NCT06483373
Title: A Single and Multiple Dose-escalation, and Food Effects of Phase I Clinical Study to Evaluate the Tolerability/Safety/Pharmacokinetics of SPH7854 Granules in Healthy Subjects.
Brief Title: A Clinical Study of SPH7854 Granules in Healthy Subjects.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPH7854-101
Record Dates: First submitted 2024-06-24; First posted 2024-07-03 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPH7854 (Experimental)
  Interventions: Drug: SPH7854
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPH7854 — SPH7854： Orally, 50-3200mg
  Arms: SPH7854
Drug: Placebo — Placebo：Orally；
  Arms: Placebo

SUMMARY:
To evaluate the safety of SPH7854 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in clinical research; Fully understand and know the study and sign the informed consent；
2. Healthy volunteers;
3. Before receiving the investigational drug, the examination results were normal or clinically insignificant;
4. Subjects who have no fertility plan/sperm donation/egg donation plan and voluntarily take effective contraceptive measures, from signing the informed consent to the prescribed time after the last dosing.

Exclusion Criteria:

1. Female subjects who are breastfeeding or have positive pregnancy results;
2. Subjects with chronic, unstable, or recurrent disease or surgery history who are judged by the investigator to be ineligible before signing informed consent;
3. Subjects suffering from allergic diseases or having a history of severe allergies;
4. Subjects who took the drug or food prohibited by the protocol prior to the first dose;
5. Subjects with evidence of infection who could not be enrolled according to the investigator's judgement;
6. Other circumstances that meet the protocol exclusion criteria.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Approximately 2 years
  Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
PK(Pharmacokinetics):Tmax | Approximately 2 years
  Time to peak plasma concentration (Tmax)
PK(Pharmacokinetics):Cmax | Approximately 2 years
  Maximum serum concentration(Cmax)
PK(Pharmacokinetics):AUC | Approximately 2 years
  Area under the plasma concentration versus time curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Sichuan University, Chengdu, China